CLINICAL TRIAL: NCT05689762
Title: Promotion of Healthy Lifestyle Habits in a Primary Care Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Varberga
Record Dates: First submitted 2022-12-23; First posted 2023-01-19 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health counselling plus E-health platform (Experimental): Receive same information as controls plus health counseling and access to E-health platform
  Interventions: Behavioral: Healthy lifestyle counseling and E-health support
- Standard care (No Intervention): Receive (1) standard care advice based on general health benefits of healthy lifestyle habits (benefits of adherence to national guidelines about physical activity and dietary habits as well as limiting alcohol intake and smoking withdrawal), (2) feedback about current lifestyle habits and health status. Tobacco users and subjects with high alcohol consumption will be referred to specialized care.

INTERVENTIONS:
Behavioral: Healthy lifestyle counseling and E-health support — Promotion of healthy lifestyle behaviors through counseling and access to E-health platform
  Arms: Health counselling plus E-health platform

SUMMARY:
Intervention aiming to promote healthy dietary and physical activity behaviors in adults with low socio-economic position in a primary health care setting

ELIGIBILITY:
Inclusion Criteria:

* age, high metabolic risk- poor lifestyle habits (diet and physical activity)

Exclusion Criteria:

* overt disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose level | Before ; at 16 weeks; at 24 months
  Blood glucose (mmol/L) assessed using chemistry kits from Ortho-Clinical Diagnostics on a Vitros-5.1 analyzer platform (Clinical Diagnostics, Raritan, NJ, United States)
Change in plasma triglycerides level | Before ; at 16 weeks; at 24 months
  Plasma triglycerides (mmol/L) : assessed using chemistry kits from Ortho-Clinical Diagnostics on a Vitros-5.1 analyzer platform (Clinical Diagnostics, Raritan, NJ, United States)

SECONDARY OUTCOMES:
Change in waist circumference | Before ; at 16 weeks; at 24 months
  waist circumference (cm) assessed by a steel tape
Change in systolic and diastolic blood pressure | Before ; at 16 weeks; at 24 months
  measured manually with a mercury sphygmomanometer
Change in HDL-cholesterol level | Before ; at 16 weeks; at 24 months
  plasma High density lipoprotein- cholesterol: assessed using chemistry kits from Ortho-Clinical

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

REFERENCES:
- [Derived] Kadi F, Nilsson A. Dynamics of Perceived Barriers to Change Physical Activity and Eating Habits in Adults Before and During a Lifestyle Intervention in a Primary Care Setting: A Mixed Methods Approach. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241273321. doi: 10.1177/21501319241273321. PMID 39148346